CLINICAL TRIAL: NCT01248793
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Golimumab in the Treatment of Chinese Subjects With Ankylosing Spondylitis
Brief Title: Study of the Safety and Efficacy of Golimumab in Chinese Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015916; C0524T29 (Other: Centocor)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Sponylitis, injection, golimumab, simponi
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Experimental)
  Interventions: Drug: Placebo; Drug: Golimumab (placebo group)
- Golimumab (Experimental)
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Placebo — Placebo subcutaneous (SC) injections at Weeks 0, 4, 8, 12, 16, and 20
  Arms: Placebo
Drug: Golimumab — Golimumab 50 mg SC injection every 4 weeks for 48 weeks
  Arms: Golimumab
Drug: Golimumab (placebo group) — Golimumab with early escape at Week 16, 50 mg SC injections at Week 24 and every 4 weeks thereafter through Week 48
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of golimumab in Chinese patients with ankylosing spondylitis

DETAILED DESCRIPTION:
Golimumab is a type of tumor necrosis factor (TNF) inhibitor. TNF is a naturally occurring substance in the body, and this substance may cause long-term inflammation. Golimumab may help fight disease by blocking the activity of TNF in the body and reducing inflammation and pain. Each patient who is allowed to join the study will be put into a group randomly, like flipping a coin. Patients may get either golimumab or placebo (which looks like the drug being studied but has no active ingredients, for example a sugar pill). The chance that the patient will get golimumab is 1 to 1, so 50% chance to receive golimumab and 50% change to receive placebo. Patients who do not have an improvement in total back pain and morning stiffness at the Week 16 visit compared to when the patients entered the study, and are in Group 1 (placebo group), will receive golimumab 50 mg every 4 weeks starting at Week 16. If the patient is in Group 2 (golimumab 50 mg), they will continue to receive golimumab every 4 weeks starting at Week 16. If the patient is in Group 1 and still receiving placebo injections, because there was improvement in total back pain at Week 16, they will receive golimumab 50 mg every 4 weeks starting from Week 24. If the patient is in Group 2 (golimumab 50 mg) or are already receiving golimumab injections at week 24, they will continue to receive golimumab every 4 weeks. Safety will be monitored throughout the study, including drawing blood and looking at laboratory tests, vital signs (eg, blood pressure), and the frequency and type of adverse events (side effects). The patient will be in the study approximately 56 weeks. Patients will receive placebo or active compound (golimumab 50 mg subcutaneous injections) every four weeks until Week 48.

ELIGIBILITY:
Inclusion Criteria:

- Have a diagnosis of definite akylosing spondylitis for at least 3 months

* Have symptoms of active disease at screening and at baseline
* no active infections

Exclusion Criteria:

* Have other inflammatory diseases that might confound the evaluations of benefit from the golimumab therapy
* Have complete ankylosis of the spine
* Have a history of latent or active granulomatous infection
* Have had a serious infection, or have been hospitalized for an infection, or have been treated with intravenous (IV) antibiotics for an infection within 2 months prior to first administration of study agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (7):
- China (7):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hefei
  - Jinan
  - Shanghai
  - Xi'an

REFERENCES:
- [Derived] Bao C, Huang F, Khan MA, Fei K, Wu Z, Han C, Hsia EC. Safety and efficacy of golimumab in Chinese patients with active ankylosing spondylitis: 1-year results of a multicentre, randomized, double-blind, placebo-controlled phase III trial. Rheumatology (Oxford). 2014 Sep;53(9):1654-63. doi: 10.1093/rheumatology/keu132. Epub 2014 Apr 11. PMID 24729398

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I: Placebo: Placebo SC injections every 4 weeks from Week 0 to Week 20(unless early escape at Week 16); Golimumab 50 mg SC injections every 4 weeks from Week 16 to Week 48 if early escape; Golimumab 50 mg SC injections every 4 weeks from Week 24 to Week 48 if not early escape
- Group II: Golimumab 50 mg: Golimumab 50 mg SC injections every 4 weeks from Week 0 to Week 48
Period: Overall Study
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg
Started | 105 | 108
Completed | 101 | 102
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Total
Number analyzed (Participants) | 105 | 108 | 213
Age Continuous [Mean (Standard Deviation); unit: years] | 30.6 (8.60) | 30.5 (10.27) | 30.5 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 87 | 90 | 177

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Ankylosing Spondylitis Response (ASAS 20) at Week 14
Description: Number of patients who achieved a >= 20% improvement in ankylosing spondylitis symptoms, including back pain, function, and inflammation
Time Frame: Week 14
Population: Intent-to-treat population according to their assigned treatment group regardless of whether or not they receive the assigned treatment
Measure: Number; unit: Participants
Groups:
- Group I: Placebo: Placebo subcutaneous (SC) injections every 4 weeks from Week 0 to Week 20 (unless early escape at Week 16); Golimumab 50 mg SC injections every 4 weeks from Week 16 to Week 20 if early escape
- Group II: Golimumab 50 mg: Golimumab 50 mg SC injections every 4 weeks from Week 0 to Week 20
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg
Number analyzed (Participants) | 105 | 108
Participants | 26 | 53

2. Secondary Outcome: Assessment of Ankylosing Spondylitis Response (ASAS 20) at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg
Number analyzed (Participants) | 105 | 108
Participants | 24 | 54

3. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 14
Description: BASFI is a participant's self-assessment, represented as a mean (Visual Analogue Scale [Score]; 0 cm [easy] to 10 cm [impossible]) of 10 questions, 8 of which relate to the participant's functional anatomy and 2 of which relate to a participant's ability to cope with everyday life. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg
Number analyzed (Participants) | 105 | 108
Score on a scale | 0.113 (2.0967) | -1.262 (2.5698)

4. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 14
Description: BASMI is a combined score of 5 components of spine flexibility, ranging from 0 (least impairment) to 10 (most impairment). A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg
Number analyzed (Participants) | 105 | 108
Score on a scale | -0.19 (0.718) | -0.42 (0.906)

ADVERSE EVENTS:
Groups:
- Placebo -> Golimumab 50 mg: Placebo SC injections every 4 weeks from Week 0 to Week 12 and early escape to receive Golimumab 50 mg SC injection every 4 weeks from Week 16 to Week 20; or Placebo SC injections every 4 weeks from Week 0 to Week 20 and crossed over to receive Golimumab 50 mg SC injections every 4 weeks from Week 24 to Week 48
- Golimumab 50 mg: Golimumab 50 mg SC injections every 4 weeks from Week 0 to Week 48
Arm/Group | Placebo -> Golimumab 50 mg | Golimumab 50 mg
Serious Adverse Events (participants affected / at risk) | 2/103 | 4/108
Other Adverse Events (participants affected / at risk) | 37/103 | 33/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo -> Golimumab 50 mg (N=103) | Golimumab 50 mg (N=108)
Uveitis (Eye disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Tuberculous Pleurisy (Infections and infestations) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo -> Golimumab 50 mg (N=103) | Golimumab 50 mg (N=108)
Upper Respiratory Tract Infection (Infections and infestations) | 23 | 24
Alanine Aminotransferase Increased (Investigations) | 7 | 7
Liver Function Test Abnormal (Investigations) | 10 | 5
Transaminases Increased (Investigations) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days